CLINICAL TRIAL: NCT04181918
Title: Action Observation Treatment and Motor Imagery as Rehabilitation Tools in Parkinson's Disease Patients
Brief Title: Action Observation Treatment in Parkinson's Patients
Acronym: AOT-PA
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Fondazione Don Carlo Gnocchi Onlus (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AOTPRFDG
Record Dates: First submitted 2019-11-18; First posted 2019-12-02 (Actual); Last update posted 2019-12-02 (Actual); Status verified 2019-05

CONDITIONS: Parkinson
Keywords: Action Observation Treatment; Motor Imagery; Randomized Controlled Study

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- AOT (Experimental): This group will observe videos depicting daily actions and afterwards they will execute the seen actions
  Interventions: Behavioral: AOT
- MI (Experimental): This group will imagine motorically the same action as the first group and afterwards they will execute the imagined actions
  Interventions: Behavioral: MI
- Control (No Intervention): This group will neither observe nor imagine actions, but simply observe videos with no motor content. Afterwards they will execute the same actions as in AOT and MI.

INTERVENTIONS:
Behavioral: AOT — During action observation, participants observe different daily actions (e.g. reading a newspaper; drinking an espresso) divided into up to four motor segments.
  Arms: AOT
Behavioral: MI — During motor imagery, participants imagine themselves performing the same daily actions as in AOT in the absence of motor output
  Arms: MI

SUMMARY:
The aim of the study is to assess the role of Action Observation Treatment (AOT) and Motor Imagery (MI) in the rehabilitation of Parkinson's disease patients, as compared to a control condition. Main outcome measures will be the results in two functional scales (FIM, UPDRS) and kinematics parameters obtained from gait analysis. Data at two months and six months follow up, respectively, will be also collected.

ELIGIBILITY:
Inclusion Criteria:

* Parkinson disease patients on Hoehn and Yahr 3-4

Exclusion Criteria:

* Mini-Mental State Examination < 24
* Fluent aphasic patients
* Apraxia
* Neglect
* major neuropsychiatric disorders

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2018-03-26 (Actual); Primary Completion 2020-03-26 (Estimated); Study Completion 2020-06-26 (Estimated)

PRIMARY OUTCOMES:
change in the functional status of the patient | Before treatment, within one week after treatment, two months' follow up
  to assess the change in the functional status of the patient, the Functional Independence Measure (FIM) will be used. FIM consists in a 7-point scale (1 = <25% independence; total assistance required, 7 = 100% independence), and it can detect changes in the patient's status in 18 categories, focusing on motor and cognitive function. Functional patients' status will assess before treatment, within one week after the end of the treatment (after treatment) and two months' follow up.
change in Parkinson disease motor symptoms | Before treatment, within one week after treatment, two months' follow up
  to assess the change in motor status of the patient, the Unified Parkinson's Disease Rating Scale (UPDRS) will be used, and it consists in a 5-point scale (0 = no signs; 4 = severe). UPDRS will be administered before treatment, within one week after the end of the treatment (after treatment) and two months' follow up.
change in kinematic parameters of the gait (velocity, footing, pace, step length) | Before treatment, within one week after treatment, two months' follow up
  to assess the change of patient's gait parameters, the kinematic analysis will be used (i.e. gait analysis). The gait analysis allows to detect fine-grain changes in kinematic parameters of the movement, through a non-invasive methodology. Gait analysis will be performed before treatment, within one week after the end of the treatment (after treatment) and two months' follow up.

CONTACTS AND LOCATIONS:
Overall Officials: Giovanni Buccino, Principal Investigator — Istituto Don Gnocchi; Claudio Rovacchi, Study Chair — Istituto Don Gnocchi
Locations (1):
- Fondazione Don Carlo Gnocchi, Parma, Italy

IPD SHARING:
Plan to Share IPD: No